CLINICAL TRIAL: NCT05600309
Title: A Phase 3 Study of MK-4280A (Coformulated Favezelimab [MK-4280] Plus Pembrolizumab [MK-3475]) Versus Standard of Care in Previously Treated Metastatic PD-L1 Positive Colorectal Cancer (KEYFORM-007)
Brief Title: A Study of Coformulated Favezelimab/Pembrolizumab (MK-4280A) Versus Standard of Care in Subjects With Previously Treated Metastatic PD-L1 Positive Colorectal Cancer (MK-4280A-007)-China Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4280A-007 China Extension; MK-4280A-007 China Extension (Other: MSD); jRCT2031210482 (Registry Identifier: jRCT(Japan Registry of Clinical Trials))
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1),; Programmed Cell Death Receptor Ligand 1 (PDL1, PD-L1); Programmed Cell Death Receptor Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Colorectal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; regorafenib; trifluridine tipiracil drug combination

STUDY DESIGN:
Masking Description: None (Open-label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Favezelimab/Pembrolizumab (Experimental): Participants will receive coformulated favezelimab/pembrolizumab (800 mg/200 mg) intravenously (IV) on Day 1, then every 3 weeks (Q3W), for up to 35 infusions.
  Interventions: Biological: favezelimab/pembrolizumab
- Standard of Care (Regorafenib or TAS-102) (Active Comparator): At the Investigator's choice, participants will receive 160 mg regorafenib orally daily on Days 1-12 of each 28-day cycle or 35 mg/m^2 TAS-102 orally twice daily on Days 1-5 and Days 8-12 of each 28-day cycle.
  Interventions: Drug: regorafenib; Drug: TAS-102

INTERVENTIONS:
Biological: favezelimab/pembrolizumab — Coformulated favezelimab/pembrolizumab (800 mg/200 mg), IV infusion
  Other Names: MK-4280A
  Arms: Favezelimab/Pembrolizumab
Drug: regorafenib — Oral
  Other Names: STIVARGA®; REGONIX®
  Arms: Standard of Care (Regorafenib or TAS-102)
Drug: TAS-102 — Oral
  Other Names: LONSURF®
  Arms: Standard of Care (Regorafenib or TAS-102)

SUMMARY:
The purpose of this China extension study is to assess the safety and efficacy of coformulated favezelimab/pembrolizumab (MK-4280A) in adult Chinese participants with metastatic colorectal cancer. The study will also compare MK-4280A with the standard of care treatment of regorafenib and TAS-102 (trifluridine and tipiracil).

The primary study hypothesis is that coformulated favezelimab/pembrolizumab (MK-4280A) is superior to standard of care with respect to overall survival.

DETAILED DESCRIPTION:
The China extension study will include participants previously enrolled in China in the global study for MK-4280A-007 (NCT05064059) plus those enrolled during the China extension enrollment period. A total of approximately 94 Chinese participants will be enrolled.

As of Amendment 3 of the supplemental statistical analysis plan, patient reported outcomes will no longer be secondary outcome measures of the study.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed colorectal adenocarcinoma that is metastatic and unresectable.
* Has measurable disease per RECIST 1.1 as assessed by the local site investigator.
* Has been previously treated for the disease and radiographically progressed on or after or could not tolerate standard treatment.
* Submits an archival (≤ 5 years) or newly obtained tumor tissue sample or newly obtained tumor tissue sample that has not been previously irradiated.
* Has an Eastern Cooperative Oncology Group Performance Score (ECOG PS) of 0 to 1 within 10 days prior to first dose of study intervention.
* Has a life expectancy of at least 3 months, based on the investigator assessment.
* Has the ability to swallow and retain oral medication and not have any clinically significant gastrointestinal abnormalities that might alter absorption.
* Has adequate organ function.

Exclusion Criteria:

* Has previously been found to have deficient mismatch repair/microsatellite instability-high (dMMR/MSI-H) tumor status.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis or leptomeningeal disease.
* Has a history of acute or chronic pancreatitis.
* Has neuromuscular disorders associated with an elevated creatine kinase (eg, inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability.
* Has urine protein greater than or equal to 1g/24h.
* A woman of childbearing potential who has a positive urine/serum pregnancy test within 24/72 hours prior to the first dose of study intervention.
* Has received prior therapy with an anti-programmed cell death 1 (PD-1), anti-programmed death ligand 1 (PD-L1), or anti-programmed cell death ligand 2 (PD-L2), anti-lymphocyte activation gene 3 (LAG-3) antibody, with a tyrosine kinase inhibitor (TKI; eg, lenvatinib) other than rapidly accelerated fibrosarcoma (RAF) inhibitors (binimetinib is permitted if combined with a RAF inhibitor), or with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4, OX-40, cluster of differentiation [CD] 137).
* Has previously received regorafenib or TAS-102.
* Has received prior systemic anticancer therapy including investigational agents within 28 days before randomization.
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy (eg, tuberculosis, known viral or bacterial infections, etc.).
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has known history of Hepatitis B or known active Hepatitis C virus infection.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2025-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (24):
- China (24):
  - The Second Affiliated Hospital of Anhui Medical University ( Site 1179), Hefei, Anhui
  - Chongqing Cancer Hospital ( Site 1151), Chongqing, Chongqing Municipality
  - Fujian Province Cancer Hospital ( Site 1178), Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center ( Site 1150), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 1154), Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University ( Site 1159), Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital ( Site 1158), Nanning, Guangxi
  - Hainan General Hospital ( Site 1177), Haikou, Hainan
  - Wuhan Union Hospital Cancer Center ( Site 1162), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 1152), Wuhan, Hubei
  - Xiangya Hospital Central South University ( Site 1171), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 1174), Changsha, Hunan
  - The Third Xiangya Hospital of Central South University ( Site 1175), Changsha, Hunan
  - Changzhou Cancer Hospital-Department of Oncology ( Site 1183), Changzhou, Jiangsu
  - Affiliated Hospital of Jiangnan University(Wuxi Fourth People's Hospital ) ( Site 1185), Wuxi, Jiangsu
  - Jilin Cancer Hospital ( Site 1163), Changchun, Jilin
  - Jinan Central Hospital ( Site 1167), Jinan, Shandong
  - Shanghai Tenth People's Hospital ( Site 1170), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center ( Site 1176), Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University ( Site 1172), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital ( Site 1161), Tianjin, Tianjin Municipality
  - Yunnan Province Cancer Hospital-Colorectal surgery ( Site 1169), Kunming, Yunnan
  - Zhejiang Cancer Hospital ( Site 1180), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital-Medical Oncology ( Site 1173), Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://trialstransparency.merckclinicaltrials.com/Study.aspx?id=4280A-007&&kw=4280A-007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 94 Chinese participants were randomized in the China extension study. Of 94 Chinese participants, 30 participants were randomized in the global portion of the MK-4280A-007 (NCT05064059) study and 64 participants were randomized in the China extension portion.
Groups:
- Favezelimab/Pembrolizumab: Participants received coformulated favezelimab/pembrolizumab (800 mg/200 mg) intravenously (IV) on Day 1, then every 3 weeks (Q3W), for up to 35 infusions.
- Standard of Care (Regorafenib or TAS-102): At the Investigator's choice, participants received 160 mg regorafenib orally daily on Days 1-12 of each 28-day cycle OR 35 mg/m^2 TAS-102 orally twice daily on Days 1-5 and Days 8-12 of each 28-day cycle.
Period: Overall Study
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Started | 50 | 44
Treated | 49 | 44
Completed | 0 | 0
Not Completed | 50 | 44
Not completed — Death | 41 | 38
Not completed — Sponsor Decision | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102) | Total
Number analyzed (Participants) | 50 | 44 | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (11.2) | 57.9 (10.4) | 56.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 14 | 37
  Male | 27 | 30 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 44 | 94
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 50 | 44 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: Up to approximately 26 months
Population: All randomized Chinese participants were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 50 | 44
Months | 9.6 [6.7 to 15.2] | 9.2 [5.6 to 14.1]
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Other; p = 0.3914, Log Rank — One-sided nominal p-value based on log-rank test; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.59 to 1.50] — HR and 95% CI were based on Cox regression model with Efron's method of tie handling with treatment as a covariate

2. Secondary Outcome: Progression-Free Survival (PFS) According Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 by BICR or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
Time Frame: Up to approximately 26 months
Population: All randomized Chinese participants were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 50 | 44
Months | 2.1 [2.1 to 2.3] | 2.1 [1.9 to 2.9]
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Other; p = 0.8091, Log Rank — One-sided nominal p-value based on log-rank test; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.78 to 1.92] — HR and 95% CI were based on Cox regression model with Efron's method of tie handling with treatment as a covariate

3. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BICR
Description: ORR was defined as the percentage of participants who achieved a confirmed complete response (CR: Disappearance of all target lesions) or partial response (PR: At least a 30% decrease in the sum of diameters of target lesion) per RECIST 1.1 as assessed by BICR
Time Frame: Up to approximately 26 months
Population: All randomized Chinese participants were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 50 | 44
Percentage of Participants | 6.0 [1.3 to 16.5] | 0.0 [0.0 to 8.0]
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Other; p = 0.0502, Miettinen & Nurminen Method — One-sided nominal p-value for testing; Difference in percentage = 6.0, 95% CI 2-sided [-2.3 to 16.3] — Difference in percentage and 95% CI were based on the Miettinen & Nurminen method

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR
Description: For participants who demonstrate confirmed CR (disappearance of all target lesions) or PR (At least a 30% decrease in the sum of diameters of target lesions), duration of response was defined as the time from the first documented evidence of CR or PR until progressive disease (PD) or death due to any cause. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions as well as an absolute increase of at least a 5 mm in the sum of diameters. The appearance of one or more new lesions was also considered PD. DOR assessments were based on blinded central imaging review with confirmation.
Time Frame: Up to approximately 26 months
Population: All randomized Chinese participants who experienced CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 3 | 0
Months | NA [NA to NA] — NA = Median, lower limit, and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. |

5. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to approximately 20 months
Population: All randomized Chinese participants who received at least one dose of study intervention were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 49 | 44
Participants | 46 | 44

6. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE is presented.
Time Frame: Up to approximately 17 months
Population: All randomized Chinese participants who received at least one dose of study intervention were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 49 | 44
Participants | 5 | 4

ADVERSE EVENTS:
Time Frame: Up to approximately 30 months
Description: Serious and Other adverse events (AEs) includes all participants who received ≥1 dose of study drug. All-Cause Mortality includes all randomized participants. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Data are reported by treatment received.
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
All-Cause Mortality (participants affected / at risk) | 41/50 | 38/44
Serious Adverse Events (participants affected / at risk) | 12/49 | 13/44
Other Adverse Events (participants affected / at risk) | 46/49 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Favezelimab/Pembrolizumab (N=49) | Standard of Care (Regorafenib or TAS-102) (N=44)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Favezelimab/Pembrolizumab (N=49) | Standard of Care (Regorafenib or TAS-102) (N=44)
Anaemia (Blood and lymphatic system disorders) | 16 (19) | 19 (20)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (6)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 9 (10) | 2 (2)
Hypothyroidism (Endocrine disorders) | 11 (12) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 4 (6)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 4 (4)
Constipation (Gastrointestinal disorders) | 4 (5) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 4 (9)
Nausea (Gastrointestinal disorders) | 3 (3) | 7 (11)
Vomiting (Gastrointestinal disorders) | 5 (8) | 4 (5)
Asthenia (General disorders) | 0 (0) | 5 (5)
Fatigue (General disorders) | 2 (2) | 3 (3)
Malaise (General disorders) | 11 (12) | 5 (5)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 3 (5) | 3 (4)
COVID-19 (Infections and infestations) | 6 (7) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Alanine aminotransferase increased (Investigations) | 10 (11) | 8 (10)
Aspartate aminotransferase increased (Investigations) | 14 (17) | 14 (16)
Blood alkaline phosphatase increased (Investigations) | 4 (6) | 6 (6)
Blood bilirubin increased (Investigations) | 6 (8) | 9 (10)
Blood lactate dehydrogenase increased (Investigations) | 5 (5) | 5 (6)
Blood thyroid stimulating hormone increased (Investigations) | 3 (3) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 7 (8) | 4 (4)
Lymphocyte count decreased (Investigations) | 2 (2) | 4 (8)
Neutrophil count decreased (Investigations) | 1 (1) | 19 (52)
Platelet count decreased (Investigations) | 3 (3) | 13 (25)
Weight decreased (Investigations) | 7 (7) | 8 (8)
White blood cell count decreased (Investigations) | 2 (2) | 17 (49)
Decreased appetite (Metabolism and nutrition disorders) | 14 (14) | 6 (6)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (5) | 5 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 (12) | 9 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6) | 3 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (10) | 2 (2)
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3)
Headache (Nervous system disorders) | 5 (5) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6) | 4 (4)
Proteinuria (Renal and urinary disorders) | 8 (8) | 11 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 8 (8)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (11)
Hypertension (Vascular disorders) | 3 (3) | 11 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT05600309/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT05600309/SAP_001.pdf